CLINICAL TRIAL: NCT06927414
Title: Exploratory Study on the Effectiveness and Safety of Light Diffraction Frame Glasses in Preventing and Controlling Myopia in Children and Adolescents
Brief Title: Light Diffraction Glasses in Preventing and Controlling Myopia in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XSKHR2024-058-006
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Myopia Progressing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light diffraction lens (Diffractive Optical Element , D.O.E) (Experimental)
  Interventions: Device: Functional lens
- H. A. L. T, highly aspheric lenslet technology (Active Comparator)
  Interventions: Device: Functional lens

INTERVENTIONS:
Device: Functional lens — Diffractive Optical Element, D.O.E, technology for controlling myopia progression in children and adolescents. and H.A.L.T, highly aspheric lenslet technology) for controlling myopia progression in children and adolescents.

SUMMARY:
This study aims to evaluate the effectiveness of lenses with light diffraction glasses in controlling the progression of myopia in children and adolescents, and to explore the feasibility of effective design, and apply personalized frame lenses for myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6-8 years old;
2. After using 1% cyclohexanone hydrochloride eye drops (Saifeijie) for ciliary muscle paralysis, binocular spherical power were within 0.00D~-1.75D, binocular cylinder power ≤ 1.50D, the anisometropia is less than 1.50D, the progression of myopia in the past year is greater than 0.5D, the best corrected far vision is at least 4.8, and the near vision is at least 5.0;
3. Within 6 months, the myopia prevention and control methods such as multifocal glasses, orthokeratology, defocusing flexible glasses, progressive glasses, atropine eye drops, red light and acupuncture and moxibustion treatment were not used;
4. The subject has a willingness to receive treatment and an informed consent form is signed by their legal guardian.

Exclusion Criteria:

1. Diagnosed constant strabismus;
2. Diagnosed pathological myopia;
3. Other congenital eye diseases;
4. Researchers believe that the patients have other reasons that are not suitable for inclusion in the project.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Subjective refraction equivalent spherical | 3 months

SECONDARY OUTCOMES:
Axial length | 3 months
Choroidal thickness | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Diseases Prevention &Treatment Center/ Shanghai Eye Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided